CLINICAL TRIAL: NCT01721369
Title: Observational Study of the Application of the ESC2009 Syncope Guidelines in Cataluña
Brief Title: Applicability of Syncope Guidelines in Cataluña
Acronym: SYNCAT
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: SYNCAT
Record Dates: First submitted 2012-06-19; First posted 2012-11-05 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2020-09

CONDITIONS: Brief Loss of Consciousness
Keywords: TLOC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transient Loss of Consciousness (T-LOC): Transient Loss of Consciousness (T-LOC). Treatment according to normal clinical practice.
  Interventions: Diagnostic Test: Transient Loss of Consciousness (T-LOC)

INTERVENTIONS:
Diagnostic Test: Transient Loss of Consciousness (T-LOC)

SUMMARY:
The aim of SYNCAT study is to study the level of adherence of the centers in Cataluña tu the Syncope Guidelines ESC2009 for the diagnosis and treatment of syncope and the impact that following them can have in the prognosis of these patients.

DETAILED DESCRIPTION:
The aim of SYNCAT study is to analyze the level of adherence of Syncope Guidelines ESC2009 for the management, diagnosis and treatment of syncope in a specific territory with similar health structure, the region of Cataluña in Spain that includes aprox. 7,000,000 inhabitants, including different complexity level of hospitals and the impact that following guidelines can have in the prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Each patient that comes from the Emergency room and/or in office doctors visit (Internal Medicine, Cardiology, Neurology...) with Transient Loss of Conscience (T-LOC)

Exclusion Criteria:

* Patients younger than 15 years old
* Pregnant women

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Transient Loss of Conscience: T-LOC
Sampling Method: Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Moya, Dr., Principal Investigator — Hospital Vall d'Hebron; Jordi Tomàs, Dr., Principal Investigator — H. Arnau de Vilanova de Lleida; Joan Nicolàs, Dr., Principal Investigator — Parc Sanitari Sant Joan de Déu; Jordi Mercè, Dr., Principal Investigator — H. Joan XXIII; Francesc Planas, Dr., Principal Investigator — H. Municipal de Badalona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Transient Loss of Consciousness (T-LOC): Patient with transient loss of consciousness (T-LOC)
Period: Overall Study
Arm/Group | Transient Loss of Consciousness (T-LOC)
Started | 581
Completed | 569
Not Completed | 12
Not completed — Not initial etiological diagnosis | 12

BASELINE CHARACTERISTICS:
Population: Patients with transient loss of consciousness (T-LOC) from the emergency service and/or external clinic visits (Cardiology, Neurology, etc).
Groups:
- Transient Loss of Consciousness (T-LOC): Patients with transient loss of consciousness (T-LOC)
Arm/Group | Transient Loss of Consciousness (T-LOC)
Number analyzed (Participants) | 581
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 214
  >=65 years | 358
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253
  Male | 328
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 581

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Adhere to the 2009 Syncope Guidelines (ESC2009)
Description: To analyze the number of patients that an etiologic diagnose was established according to the New Syncope Guidelines ESC2009 in the hospital care, in a particular community with hospitals with different levels of care in a specific region of Spain.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Transient Loss of Consciousness (T-LOC)
Number analyzed (Participants) | 569
Participants | 233

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious adverse events (SAE) were recollect at 1 year follow up, other adverse events were not recollected in this observational study.
Arm/Group | Transient Loss of Consciousness (T-LOC)
Serious Adverse Events (participants affected / at risk) | 163/569
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transient Loss of Consciousness (T-LOC) (N=569)
Life-threatening illness or injury (General disorders) | 4
Hospitalization (General disorders) | 123
Permanent insufficiency of a body structure or a body function (General disorders) | 1
Death (General disorders) | 35

LIMITATIONS AND CAVEATS:
Observational study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No